CLINICAL TRIAL: NCT00982111
Title: A Randomized, Multicenter, Open-Label Phase 3 Study of Pemetrexed-Cisplatin Chemotherapy Plus Necitumumab (IMC-11F8) Versus Pemetrexed-Cisplatin Chemotherapy Alone in the First-Line Treatment of Patients With Stage IV Nonsquamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: First-line Treatment of Patients With Stage IV Nonsquamous Non-Small Cell Lung Cancer With Necitumumab (IMC-11F8) and Pemetrexed-Cisplatin
Acronym: INSPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Quintiles, Inc. (Industry); Parexel (Industry); PPD Development, LP (Industry); Medidata Solutions (Industry); Laboratory Corporation of America (Industry); University of Colorado, Denver (Other); Thermo Fisher Scientific, Inc (Industry); Pacific Biomarkers (Other); Intertek (Industry); Sysmex Inostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13908; 2009-012574-12 (EudraCT Number); CP11-0805 (Other: ImClone Systems); I4X-IE-JFCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Nonsquamous; Non Small Cell Lung Cancer; First line treatment; Monoclonal; Antibodies; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Necitumumab + Pemetrexed + Cisplatin (Experimental): Necitumumab + Pemetrexed + Cisplatin
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Biological: Necitumumab
- Pemetrexed + Cisplatin (Active Comparator): Pemetrexed + Cisplatin
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 milligram per square meter (mg/m2) administered Intravenously (I.V.) on Day 1 of every 3-week cycle, for a maximum of six cycles
  Other Names: Alimta®; LY231514
Drug: Cisplatin — 75 mg/m2 administered I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
Biological: Necitumumab — 800 mg (absolute dose) on Days 1 and 8 of every 3-week cycle, administered as an I.V.
  Other Names: IMC-11F8; LY3012211; Portrazza®
  Arms: Necitumumab + Pemetrexed + Cisplatin

SUMMARY:
The research study is testing the investigational drug necitumumab in the treatment of advanced non-small cell lung cancer. The aim of this study is to determine if necitumumab, given together with a standard chemotherapy combination consisting of cisplatin and pemetrexed will be more effective in improving participant disease than the standard chemotherapy combination alone.

DETAILED DESCRIPTION:
Multinational, randomized, multicenter, open-label Phase 3 study of 633 participants with advanced, nonsquamous (Stage IV) NSCLC. Participants will be randomized on a 1:1 basis to receive first-line necitumumab plus chemotherapy consisting of pemetrexed and cisplatin in study Arm A, or first-line pemetrexed-cisplatin chemotherapy alone in Arm B.

Baseline radiographic assessment of disease will be performed within 21 days prior to randomization (first treatment will be administered within 7 days following randomization).

Participants will undergo radiographic assessment (computed tomography or magnetic resonance imaging) of disease status every 6 weeks (± 3 days), until there is radiographic documentation of progressive disease (PD). Chemotherapy will continue for a maximum of six cycles in each arm (Or until there is radiographic documentation of PD, toxicity requiring cessation, protocol noncompliance or withdrawal of consent); participants in Arm A only will continue to receive necitumumab until there is radiographic documentation of PD, toxicity requiring cessation, protocol noncompliance, or withdrawal of consent.

After the end-of-study-visit (following PD), follow-up information regarding further anticancer treatment and survival will be collected every 2 months (± 7 days). For participants who discontinue study for reasons other than PD (eg, symptomatic deterioration), information on disease progression will also be collected until PD is documented. Follow-up will continue as long as the participant is alive, or until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed nonsquamous (adenocarcinoma/large cell or other) non small cell lung cancer
* Has Stage IV disease at the time of study entry
* Measurable or nonmeasurable disease (as defined by the Response Evaluation Criteria in Solid Tumors RECIST 1.0) at the time of study entry (participants with only truly nonmeasurable disease are not eligible)
* Has resolution to Grade ≤ 1 of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (with the exception of alopecia)
* Has an Eastern Cooperative Oncology Group performance status score of 0-2
* Has adequate hepatic function
* Has adequate renal function
* Has adequate hematologic function
* If female, is surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method during and for 6 months after the treatment period (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method). If male, the participants surgically sterile or compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period
* Female participants of childbearing potential must have a negative serum

Exclusion Criteria:

* Has squamous non small cell lung cancer
* Has received prior anticancer therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the Epidermal Growth Factor Hormone (EGFR), vascular endothelial growth factor (VEGF), or VEGF receptor
* Received previous chemotherapy for advanced NSCLC (participants who have received adjuvant chemotherapy are eligible if the last administration of the prior adjuvant regimen occurred at least 1 year prior to randomization)
* Undergone major surgery or received any investigational therapy in the 4 weeks prior to randomization
* Undergone chest irradiation within 12 weeks prior to randomization (except palliative irradiation of bone lesions, which is allowed)
* Has brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants. Participants who have undergone previous radiotherapy for brain metastases, who are now nonsymptomatic and no longer require treatment with steroids or anticonvulsants, are eligible
* Has superior vena cava syndrome contraindicating hydration
* Has current clinically-relevant coronary artery disease or uncontrolled congestive heart failure
* Has experienced myocardial infarction within 6 months prior to randomization
* Has an ongoing or active infection (requiring antibiotics), including active tuberculosis or known infection with the human immunodeficiency virus
* Has a history of significant neurological or psychiatric disorders, including dementia, seizures, or bipolar disorder, potentially precluding protocol compliance
* Has Grade ≥ 2 peripheral neuropathy
* Has significant third space fluid retention, requiring repeated drainage
* Has any other serious uncontrolled medical disorders or psychological conditions that would, in the opinion of the investigator, limit the participant's ability to complete the study or sign an informed consent document The participant has a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of IMC-11F8, or any other contraindication to one of the administered treatments
* Is pregnant or breastfeeding
* Has a known history of drug abuse
* Has a concurrent active malignancy other than adequately-treated basal cell carcinoma of the skin or preinvasive carcinoma of the cervix. A participant with previous history of malignancy other than NSCLC is eligible, provided that he/she has been free of disease for ≥ 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2009-11-02 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (94):
- ImClone Investigational Site, Nyack, New York, United States
- Australia (3):
  - ImClone Investigational Site, Kogarah, New South Wales
  - ImClone Investigational Site, Hobart, Tasmania
  - ImClone Investigational Site, East Bentleigh, Victoria
- Austria (2):
  - ImClone Investigational Site, Rankweil
  - ImClone Investigational Site, Vienna
- Belgium (3):
  - ImClone Investigational Site, Duffel
  - ImClone Investigational Site, Liège
  - ImClone Investigational Site, Namur
- Brazil (11):
  - ImClone Investigational Site, Barretos - SP
  - ImClone Investigational Site, Brasilia, Distrito Federal
  - ImClone Investigational Site, Goiania - GO
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Itajaí
  - ImClone Investigational Site, Lajeado
  - ImClone Investigational Site, Porto Alegre/RS
  - ImClone Investigational Site, Ribeirão Preto - SP
  - ImClone Investigational Site, Salvador
  - ImClone Investigational Site, Santo Andre - SP
  - ImClone Investigational Site, São Paulo - SP
- ImClone Investigational Site, Montreal, Quebec, Canada
- ImClone Investigational Site, Pula, Croatia
- France (2):
  - ImClone Investigational Site, Caen
  - ImClone Investigational Site, Paris
- Germany (18):
  - ImClone Investigational Site, Berlin
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Frankfurt
  - ImClone Investigational Site, Gauting
  - ImClone Investigational Site, Großhansdorf
  - ImClone Investigational Site, Halle
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Heidelberg
  - ImClone Investigational Site, Hemer
  - ImClone Investigational Site, Hofheim
  - ImClone Investigational Site, Karlsruhe
  - ImClone Investigational Site, Lostau
  - ImClone Investigational Site, Löwenstein
  - ImClone Investigational Site, Mainz
  - ImClone Investigational Site, München
  - ImClone Investigational Site, Münster
  - ImClone Investigational Site, Regensburg
  - ImClone Investigational Site, Ulm
- Greece (3):
  - ImClone Investigational Site, Athens
  - ImClone Investigational Site, Heraklion, Crete
  - ImClone Investigational Site, Pátrai
- Hungary (6):
  - ImClone Investigational Site, Budapest
  - ImClone Investigational Site, Deszk
  - ImClone Investigational Site, Mosonmagyaróvár
  - ImClone Investigational Site, Székesfehérvár
  - ImClone Investigational Site, Szombathely
  - ImClone Investigational Site, Törökbálint
- Italy (7):
  - ImClone Investigational Site, Lido di Camaiore, Lucca
  - ImClone Investigational Site, Aviano, Pordenone
  - ImClone Investigational Site, Frosinone
  - ImClone Investigational Site, Genova
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Parma
  - ImClone Investigational Site, Perugia
- Poland (6):
  - ImClone Investigational Site, Olsztyn
  - ImClone Investigational Site, Otwock
  - ImClone Investigational Site, Poznan
  - ImClone Investigational Site, Radom
  - ImClone Investigational Site, Szczecin
  - ImClone Investigational Site, Wroclaw
- Portugal (2):
  - ImClone Investigational Site, Coimbra
  - ImClone Investigational Site, Lisbon
- Romania (6):
  - ImClone Investigational Site, Brasov
  - ImClone Investigational Site, Bucharest
  - ImClone Investigational Site, Cluj-Napoca
  - ImClone Investigational Site, Craiova, Dolj
  - ImClone Investigational Site, Iași
  - ImClone Investigational Site, Sibiu
- Russia (6):
  - ImClone Investigational Site, Ivanovo
  - ImClone Investigational Site, Kirov
  - ImClone Investigational Site, Omsk
  - ImClone Investigational Site, Saint Petersburg
  - ImClone Investigational Site, Ufa
  - ImClone Investigational Site, Yaroslavi
- Slovakia (2):
  - ImClone Investigational Site, Bratislava
  - ImClone Investigational Site, Nitra
- South Africa (2):
  - ImClone Investigational Site, Bloemfontein, Free State
  - ImClone Investigational Site, Pretoria, Gauteng
- Spain (6):
  - Imclone Investigational Site, Seville, Andalusia
  - ImClone Investigational Site, Barcelona, Catalonia
  - ImClone Investigational Site, Terrassa, Catalonia
  - ImClone Investigational Site, Madrid, Communidad de Madrid
  - ImClone Investigational Site, Majadahonda, Communidad de Madrid
  - ImClone Investigational Site, L'Hospitalet de Llobregat
- United Kingdom (6):
  - ImClone Investigational Site, Aberdeen
  - ImClone Investigational Site, Bournemouth
  - ImClone Investigational Site, Edinburgh
  - ImClone Investigational Site, Guildford
  - ImClone Investigational Site, Leeds
  - ImClone Investigational Site, Preston

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and assigned data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Paz-Ares L, Mezger J, Ciuleanu TE, Fischer JR, von Pawel J, Provencio M, Kazarnowicz A, Losonczy G, de Castro G Jr, Szczesna A, Crino L, Reck M, Ramlau R, Ulsperger E, Schumann C, Miziara JE, Lessa AE, Dediu M, Balint B, Depenbrock H, Soldatenkova V, Kurek R, Hirsch FR, Thatcher N, Socinski MA; INSPIRE investigators. Necitumumab plus pemetrexed and cisplatin as first-line therapy in patients with stage IV non-squamous non-small-cell lung cancer (INSPIRE): an open-label, randomised, controlled phase 3 study. Lancet Oncol. 2015 Mar;16(3):328-37. doi: 10.1016/S1470-2045(15)70046-X. Epub 2015 Feb 18. PMID 25701171

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause and participants who were alive and on study at conclusion however were off treatment.
Groups:
- Necitumumab + Pemetrexed + Cisplatin: Necitumumab + Pemetrexed + Cisplatin
  Necitumumab: 800 milligrams (mg) (absolute dose) on Days 1 and 8 of every 3-week cycle.
  Pemetrexed: 500 mg/square meter (mg/m2) intravenous (I.V.) on Day 1 of every 3-week cycle, for a maximum of six cycles.
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles.
- Pemetrexed + Cisplatin: Pemetrexed + Cisplatin
  Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles.
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles.
Period: Overall Study
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Started | 315 | 318
Received at Least 1 Dose of Study Drug | 304 | 312
Death Due to Any Cause | 236 | 246
Completed | 236 | 246
Not Completed | 79 | 72
Not completed — Adverse Event | 1 | 1
Not completed — Progressive Disease | 46 | 39
Not completed — Lost to Follow-up | 9 | 6
Not completed — New Anti-Cancer Therapy | 5 | 5
Not completed — Medical Decision | 1 | 0
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Global Study End | 0 | 1
Not completed — Sponsor's Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Necitumumab + Pemetrexed + Cisplatin: Necitumumab: 800 mg (absolute dose) on Days 1 and 8 of every 3-week cycle, administered as an I.V. infusion
  Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
- Pemetrexed + Cisplatin: Pemetrexed + Cisplatin
  Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
- Total: Total of all reporting groups
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin | Total
Number analyzed (Participants) | 315 | 318 | 633
Age, Customized [Median (Full Range); unit: years] | 61.0 [26 to 84] | 60.0 [34 to 88] | 61.00 [26 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 108 | 209
  Male | 214 | 210 | 424
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 46 | 93
  Not Hispanic or Latino | 268 | 272 | 540
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 292 | 298 | 590
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 16 | 13 | 29
  Romania | 21 | 31 | 52
  Hungary | 23 | 22 | 45
  United States | 0 | 1 | 1
  United Kingdom | 11 | 11 | 22
  Portugal | 6 | 1 | 7
  Spain | 40 | 27 | 67
  Greece | 5 | 10 | 15
  Canada | 2 | 1 | 3
  Austria | 8 | 11 | 19
  Belgium | 8 | 9 | 17
  Brazil | 37 | 35 | 72
  Poland | 28 | 24 | 52
  Italy | 17 | 19 | 36
  South Africa | 2 | 5 | 7
  Slovakia | 3 | 1 | 4
  Australia | 6 | 8 | 14
  France | 7 | 3 | 10
  Germany | 75 | 84 | 159
  Croatia | 0 | 2 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Number; unit: participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). 0 - Fully Active. 1 - Ambulatory, Restricted Strenuous Activity. 2 - Ambulatory, No Work Activities. 3 - Partially Confined to Bed, Limited Self Care. 4 - Completely Disabled. 5 - Death.
  participants
    0 | 115 | 132 | 247
    1 | 183 | 166 | 349
    2 | 16 | 20 | 36
    Missing | 1 | 0 | 1
Smoking [Number; unit: participants]
  Ex-Light Smoker | 26 | 27 | 53
  Nonsmoker | 51 | 53 | 104
  Smoker | 238 | 238 | 476
Disease Stage at Study Entry [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes. Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  participants
    Stage IIIB | 9 | 11 | 20
    Stage IV | 305 | 307 | 612
    Missing | 1 | 0 | 1
Disease Histology [Number; unit: participants]
  Adenocarcinoma/Large Cell Carcinoma | 307 | 311 | 618
  Other | 7 | 7 | 14
  Missing | 1 | 0 | 1
Sites of Metastatic Disease [Number; unit: participants] — Participants may record multiple sites of metastatic disease.
  participants
    Bone | 103 | 109 | 212
    Brain | 27 | 25 | 52
    Liver | 58 | 64 | 122
    Lung | 259 | 268 | 527
    Lymph Nodes | 239 | 240 | 479
    Peritoneal | 21 | 22 | 43
    Pleural | 111 | 111 | 222
    Skin | 7 | 5 | 12
    Soft Tissue | 19 | 21 | 40
    Other | 87 | 93 | 180

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time (OS)
Description: OS is defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive. OS was estimated using the Kaplan-Meier method.
Time Frame: Randomization to Death from Any Cause (Up to 31.6 Months)
Population: All randomized participants. Censored participants: Necitumumab + Pemetrexed + Cisplatin =79, Pemetrexed + Cisplatin=72
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Necitumumab + Pemetrexed + Cisplatin: Necitumumab + Pemetrexed + Cisplatin
  Necitumumab: 800 mg (absolute dose) on Days 1 and 8 of every 3-week cycle, administered as an I.V. infusion
  Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 315 | 318
Months | 11.3 [9.5 to 13.4] | 11.5 [10.1 to 13.1]
Statistical Analysis 1: Comparison: Necitumumab + Pemetrexed + Cisplatin vs Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.9561, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.21]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization until the first radiographic documentation of measured progressive disease as defined by RECIST (Version 1.0), or death from any cause. Participants who die without a reported prior progression will be considered to have progressed on the day of their death. Participants who did not progress or were lost to follow-up were censored at the day of their last radiographic tumor assessment. If no baseline or postbaseline radiologic assessment was available, the participant was censored at the date of randomization. If death or PD occurs after two or more consecutive missing radiographic visits, censoring occurred at the date of the last radiographic visit prior to the missed visits.
Time Frame: Randomization to Measured Progressive Disease or Death from Any Cause (Up to 30.4 Months)
Population: All randomized participants. Censored participants: Necitumumab + Pemetrexed + Cisplatin=84, Pemetrexed + Cisplatin=79
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 315 | 318
Months | 5.6 [5.1 to 6.0] | 5.6 [4.8 to 5.7]
Statistical Analysis 1: Comparison: Necitumumab + Pemetrexed + Cisplatin vs Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.6647, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.80 to 1.16]

3. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) (Objective Tumor Response Rate [ORR])
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.0, CR was defined as the disappearance of all target and non-target lesions; PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD. Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence)/total number of participants treated) * 100.
Time Frame: Baseline to Measured Progressive Disease (Up to 30.4 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 315 | 318
percentage of participants | 31.1 [26.3 to 36.4] | 32.1 [27.2 to 37.4]
Statistical Analysis 1: Comparison: Necitumumab + Pemetrexed + Cisplatin vs Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.7945, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.68 to 1.34]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from study enrollment/randomization to the first observation of measured progressive disease, death from any cause, or early discontinuation of treatment or initiation of new anti-cancer therapies. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Progressive Disease (PD) was defined as having at least a 20% increase in sum of longest diameter of target lesions. Time to treatment failure was censored at the date of the last follow-up visit for participants who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: Randomization to Measured Progressive Disease, Death from Any Cause, Discontinuation of Treatment or Initiation of New Anticancer Therapy (Up to 30.4 Months)
Population: All randomized participants. Censored participants: Necitumumab + Pemetrexed + Cisplatin = 10, Pemetrexed + Cisplatin = 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 315 | 318
Months | 3.5 [3.2 to 3.9] | 4.3 [3.3 to 4.8]
Statistical Analysis 1: Comparison: Necitumumab + Pemetrexed + Cisplatin vs Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.0459, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [1.00 to 1.39]

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab
Time Frame: Predose Day 1 of Cycle 2,3,4,5 and 6 Prior to Necitumumab Infusion, Up to 23 Weeks
Population: Participants who were randomized to necitumumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/ml)
Arm/Group | Necitumumab + Pemetrexed + Cisplatin
Number analyzed (Participants) | 315
micrograms/milliliter (ug/ml)
  Predose Cycle 2 Day 1: number analyzed (Participants) | 222
  Predose Cycle 2 Day 1 | 57.5 (84.5)
  Predose Cycle 3 Day 1: number analyzed (Participants) | 185
  Predose Cycle 3 Day 1 | 80.8 (89.3)
  Predose Cycle 4 Day 1: number analyzed (Participants) | 159
  Predose Cycle 4 Day 1 | 110 (82.9)
  Predose Cycle 5 Day 1: number analyzed (Participants) | 131
  Predose Cycle 5 Day 1 | 115 (81.8)
  Predose Cycle 6 Day 1: number analyzed (Participants) | 110
  Predose Cycle 6 Day 1 | 119 (68.9)

6. Secondary Outcome: Number of Participants With Serum Anti-Necitumumab Antibody Assessment (Immunogenicity)
Description: A participant was considered to have an anti-Necitumumab antibody response if anti-drug antibodies (ADA) were confirmed positive. Treatment emergent antibodies were defined as any anti-Necitumumab antibody titer equal to or greater than 4-fold the participant's baseline titer.
Time Frame: Baseline to Study Completion (Up to 31.6 Months)
Population: All randomized participants who received at least one dose of necitumumab and had evaluable antibody data.
Measure: Number; unit: participants
Groups:
- Necitumumab + Pemextrexed + Cisplatin: Necitumumab + Pemetrexed + Cisplatin
  Necitumumab: 800 mg (absolute dose) on Days 1 and 8 of every 3-week cycle, administered as an I.V. infusion
  Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
  Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
Arm/Group | Necitumumab + Pemextrexed + Cisplatin
Number analyzed (Participants) | 301
participants
  1 Positive Titer | 37
  Antibodies Detected | 18

7. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcomes (PRO) Using the European Quality of Life-5 Dimensions (EQ-5D)
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three level scale 1-3 (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension).
Time Frame: Baseline, Cycle 6 (Cycle = 3 weeks)
Population: All randomized participants who had evaluable baseline and postbaseline EQ-5D data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 143 | 147
units on a scale | 0.0419 (0.28230) | 0.0478 (0.22645)

8. Secondary Outcome: Mean Change From Baseline in PRO as Measured Using the Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 items: 6 items focused on lung cancer symptoms [loss of appetite, fatigue, cough, dyspnea (shortness of breath), hemoptysis (blood in sputum), and pain] and 3 items were global items (symptom distress, interference with activity level, and global quality of life). Participant responses to each item were measured using visual analogue scales (VAS) with 100-mm lines. A higher score for any item represented a higher level of symptoms/problems. Scores for each of the reported categories ranged from 0 (for best outcome) to 100 (for worst outcome). The Average Symptom Burden Index (ASBI) was the mean of the 6 symptom items of the LCSS, and the Total LCSS was the mean of all 9 LCSS items. ASBI and Total LCSS were not computed for a participant if he/she had 1 or more missing values for the 6 and 9 items, respectively.
Time Frame: Baseline, Cycle 6 (Cycle =3 Weeks)
Population: All randomized participants who had evaluable baseline and postbaseline LCSS data.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 315 | 318
millimeter (mm)
  Loss of Appetite: number analyzed (Participants) | 142 | 147
  Loss of Appetite | 4.6 (46.18) | 0.6 (27.52)
  Fatigue: number analyzed (Participants) | 142 | 148
  Fatigue | 4.5 (31.24) | 1.6 (28.75)
  Cough: number analyzed (Participants) | 143 | 148
  Cough | -9.1 (31.08) | -10.3 (27.88)
  Dyspnea: number analyzed (Participants) | 141 | 146
  Dyspnea | -2.8 (26.32) | -1.5 (23.67)
  Hemoptysis: number analyzed (Participants) | 141 | 147
  Hemoptysis | -1.1 (11.92) | -1.1 (7.81)
  Pain: number analyzed (Participants) | 142 | 147
  Pain | -4.2 (27.22) | -7.1 (26.64)
  Overall Symptoms: number analyzed (Participants) | 141 | 146
  Overall Symptoms | -3.1 (31.22) | -7.4 (27.11)
  Quality of Life: number analyzed (Participants) | 142 | 146
  Quality of Life | 2.5 (26.01) | -3.3 (24.91)
  Interference: number analyzed (Participants) | 141 | 145
  Interference | 3.2 (27.15) | -4.0 (31.39)
  Average Symptom Burden Index (ASBI): number analyzed (Participants) | 133 | 138
  Average Symptom Burden Index (ASBI) | -0.9 (18.35) | -3.1 (13.11)
  LCSS Total Score: number analyzed (Participants) | 132 | 132
  LCSS Total Score | 0.1 (17.59) | -4.3 (13.90)

9. Secondary Outcome: Epidermal Growth Factor Hormone (EGFR) Protein Expression Measured by Immunohistochemistry (IHC)
Description: EGFR IHC H-score = weighted sum of % 1+ cells, twice % 2+ cells, and three times % 3+ cells. IHC H-score criteria assesses participants with a low EGFR expression defined by a H-score cutoff value of < 200 and participants with a high EGFR expression defined by a H-score of cutoff value of >=200.
Time Frame: Baseline
Population: Translational research population included all participants who: (1) received at least one dose of study drug; (2) had a valid non-missing result for EGFR H-Score; and (3) were enrolled for more than 2 cycles prior to the decision to terminate enrollment.
Measure: Mean (Standard Deviation); unit: H-Score
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 245 | 245
H-Score
  H-score <200: number analyzed (Participants) | 144 | 146
  H-score <200 | 69.06 (64.68) | 66.23 (64.15)
  H-score >=200: number analyzed (Participants) | 101 | 99
  H-score >=200 | 259.35 (27.65) | 256.26 (29.10)

10. Secondary Outcome: Percentage of Participants With EGFR Measured by IHC
Description: as for outcome 9
Time Frame: Baseline
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Necitumumab + Pemetrexed + Cisplatin | Pemetrexed + Cisplatin
Number analyzed (Participants) | 245 | 245
percentage of participants
  H-score <200: number analyzed (Participants) | 144 | 146
  H-score <200 | 58.8 | 59.6
  H-score >=200: number analyzed (Participants) | 101 | 99
  H-score >=200 | 41.2 | 40.4

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly
Groups:
- Necitumumab+Pemetrexed+Cisplatin: Necitumumab + Pemetrexed + Cisplatin Necitumumab: 800 mg (absolute dose) on Days 1 and 8 of every 3-week cycle Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
- Pemetrexed+Cisplatin: Pemetrexed + Cisplatin Pemetrexed: 500 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles Cisplatin: 75 mg/m2 I.V. on Day 1 of every 3-week cycle, for a maximum of six cycles
Arm/Group | Necitumumab+Pemetrexed+Cisplatin | Pemetrexed+Cisplatin
All-Cause Mortality (participants affected / at risk) | 236/304 | 246/312
Serious Adverse Events (participants affected / at risk) | 158/304 | 130/312
Other Adverse Events (participants affected / at risk) | 296/304 | 303/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab+Pemetrexed+Cisplatin (N=304) | Pemetrexed+Cisplatin (N=312)
Anaemia (Blood and lymphatic system disorders) | 12 (15) | 13 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (9) | 5 (6)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (12) | 6 (6)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (4)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (10) | 7 (7)
Asthenia (General disorders) | 8 (11) | 2 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 8 (10) | 7 (7)
General physical health deterioration (General disorders) | 6 (7) | 4 (5)
Mucosal inflammation (General disorders) | 4 (4) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Intestinal gangrene (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (2)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (14) | 6 (7)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 5 (8)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 10 (10)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 4 (5)
Convulsion (Nervous system disorders) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 2 (2)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (5) | 6 (7)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Analgesic therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Superior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Necitumumab+Pemetrexed+Cisplatin (N=304) | Pemetrexed+Cisplatin (N=312)
Anaemia (Blood and lymphatic system disorders) | 72 (155) | 91 (200)
Leukopenia (Blood and lymphatic system disorders) | 45 (92) | 36 (61)
Lymphopenia (Blood and lymphatic system disorders) | 16 (53) | 17 (26)
Neutropenia (Blood and lymphatic system disorders) | 92 (179) | 99 (217)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (43) | 23 (42)
Tinnitus (Ear and labyrinth disorders) | 15 (18) | 16 (18)
Conjunctivitis (Eye disorders) | 31 (46) | 6 (6)
Lacrimation increased (Eye disorders) | 4 (4) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 19 (25) | 15 (15)
Abdominal pain upper (Gastrointestinal disorders) | 26 (36) | 25 (29)
Constipation (Gastrointestinal disorders) | 91 (133) | 83 (124)
Diarrhoea (Gastrointestinal disorders) | 90 (148) | 51 (78)
Dyspepsia (Gastrointestinal disorders) | 16 (21) | 18 (28)
Nausea (Gastrointestinal disorders) | 174 (392) | 183 (403)
Stomatitis (Gastrointestinal disorders) | 30 (41) | 12 (22)
Vomiting (Gastrointestinal disorders) | 105 (213) | 104 (180)
Asthenia (General disorders) | 88 (192) | 68 (146)
Fatigue (General disorders) | 87 (164) | 95 (171)
Mucosal inflammation (General disorders) | 50 (104) | 27 (36)
Non-cardiac chest pain (General disorders) | 11 (16) | 16 (22)
Oedema peripheral (General disorders) | 40 (52) | 41 (51)
Pyrexia (General disorders) | 46 (57) | 22 (32)
Oral candidiasis (Infections and infestations) | 18 (22) | 5 (5)
Paronychia (Infections and infestations) | 28 (67) | 0 (0)
Urinary tract infection (Infections and infestations) | 19 (21) | 16 (21)
Blood creatinine increased (Investigations) | 21 (34) | 18 (23)
Weight decreased (Investigations) | 39 (53) | 24 (28)
Anorexia (Metabolism and nutrition disorders) | 110 (174) | 97 (171)
Fluid retention (Metabolism and nutrition disorders) | 17 (39) | 12 (22)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (34) | 10 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 30 (51) | 13 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (34) | 23 (33)
Hypomagnesaemia (Metabolism and nutrition disorders) | 75 (185) | 36 (66)
Hyponatraemia (Metabolism and nutrition disorders) | 23 (36) | 20 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (40) | 20 (24)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 (26) | 15 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (22) | 17 (19)
Dizziness (Nervous system disorders) | 38 (52) | 26 (37)
Dysgeusia (Nervous system disorders) | 21 (27) | 32 (43)
Headache (Nervous system disorders) | 30 (41) | 27 (32)
Paraesthesia (Nervous system disorders) | 16 (20) | 8 (9)
Depression (Psychiatric disorders) | 18 (20) | 10 (11)
Insomnia (Psychiatric disorders) | 17 (23) | 15 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (75) | 48 (59)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (62) | 41 (52)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 10 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (31) | 18 (20)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 42 (119) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 43 (62) | 11 (13)
Hirsutism (Skin and subcutaneous tissue disorders) | 5/95 (5) | 0/107 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (48) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 125 (346) | 20 (23)
Rash generalised (Skin and subcutaneous tissue disorders) | 28 (62) | 5 (5)
Hypertension (Vascular disorders) | 17 (24) | 29 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days